CLINICAL TRIAL: NCT06754982
Title: Temporal Differences in Pain, Muscle Stiffness, and Function in Subjects With Plantar Fasciitis After Myofascial Release Therapy
Acronym: TDPSFPFMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Ignacio Gajardo Valenzuela, Principal Investigator, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N°116/2023
Record Dates: First submitted 2024-11-15; First posted 2025-01-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Plantar Fasciitis of Both Feet
Keywords: Plantar fasciitis; Myofascial release; manual therapy
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: A randomized, two-group parallel equivalence clinical trial will be conducted. Participants will be randomly assigned to one of two groups, 15 minutes of myofascial release, 30 minutes of myofascial release. In order to establish equivalence between groups, the equivalence limit or tolerance range will be adopted so that the groups do not present more than half of the value of the main variable that can be used in a superiority test (12). Therefore, for this research the adopted value will be 0.65 kg/cm2 in the pressure pain threshold, because an average change of 1.3 kg/cm2 has been observed.(10) Randomization and evaluations will be carried out by external assistants.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 15 minutes (Experimental): The group will receive 15 minutes of myofascial release. Each intervention will be performed only on the affected limb. 9 myofascial release techniques will be applied to each group, each procedure will last 1 minute and 40 seconds.
  Interventions: Other: Myofascial release
- Gruops 30 minutes (Experimental): The group will receive 30 minutes of myofascial release. Each intervention will be performed only on the affected limb. Nine myofascial release techniques will be applied to each group, each procedure will last 3 minutes and 20 seconds.
  Interventions: Other: Myofascial release

INTERVENTIONS:
Other: Myofascial release — Nine myofascial release techniques will be applied to each group: Transverse hamstring play; Transverse hamstring and adductor magnus play: posterior to anterior pressure; Transverse gastrocnemius-soleus play; Tibia bone clearing: posterior tibia; Tibia bone clearing: prone grip with half chisel; Lateral fascial distraction of the tibia; Lateral elongation of the peroneal tissue; Cross-friction of the gastrocnemius-soleus musculotendinous junction; Manipulation of the plantar fascia.

SUMMARY:
Plantar fasciitis (PF) is a common condition in the population. One of the interventions used to resolve this condition is myofascial release (MR), which consists of massages that help reduce pain and increase mobility. MR has shown efficacy when applied for 30 minutes, however, it is necessary to compare it with a 15-minute MR intervention, since in clinical practice optimizing time is essential. Accordingly, the present research seeks to evaluate whether there are differences in the application time of myofascial release in people with PF.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is an acute inflammation of the fascia resulting from degenerative irritation from the median tuberosity of the heel bone to surrounding perifascial structures. Histological findings include granulation tissue, microtears, collagen disorders, and in particular a lack of normal inflammation. It is one of the most common causes of musculoskeletal pain, with a population prevalence in adults aged 50 years or older of 9.6% (95% CI: 8.8 to 10.5) and a population prevalence of disabling pain of 7.9% (95% CI: 7.1 to 8.7), slightly more present in women than in men, with a history of knee, hip, and back pain. It is characterized by pain on the first step and pain during weight-bearing tasks, particularly after periods of rest. Among the possible low-cost and noninvasive treatments that have shown efficacy Manual therapy (MT) is a popular treatment for PF. TM includes treatments such as joint and soft tissue mobilizations, manipulations, myofascial trigger point release, and stretch-contraction-relaxation. In particular, myofascial release is a gradual soft tissue stretching by the clinician that is guided entirely by feedback from the recipient's body to determine the direction, strength, and duration of the stretch to address specific soft tissue restrictions.

TM has been frequently used to treat PF, systematic reviews have reported positive results on pain, function, and pressure pain threshold, but suggest that they should be viewed with caution due to poor methodological quality, intervention heterogeneity in dosing (frequency, intensity, and duration), techniques, and outcome measures, and the frequent use of secondary manual therapy co-interventions. The application of myofascial release is varied in the number of procedures, application time of each technique and total application time of the intervention, without a clear justification regarding the decision of each of these options. A clinical trial applied a protocol for 4 weeks, where each session was performed in 30 minutes, and demonstrated that myofascial release is more effective than the control group, presenting a change in the average pressure pain threshold of 1.3 kg/cm2 at the end of the 4-week treatment. This change is considered clinically important, given that in the literature it has been reported that this difference is > 1.16 kg/cm2. However, the reason for the time used, the number of techniques and the choice of techniques is not justified. In addition, there are no investigations in the literature on the specific effect of myofascial release with a shorter application time in PF. On the other hand, studies with deep massage, a manual therapy technique, combined with flexibility exercise has proven to be effective with an execution time of 10 minutes. Under this context and considering that in clinical practice the optimization of times is essential, it is relevant to carry out a clinical equivalence trial that allows to determine the efficacy of isolated myofascial release in PF, with a 30-minute intervention protocol already carried out and that demonstrated positive effects on the pressure pain threshold, contrasted with a time of less than 15 minutes. Given the context raised, the question arises: In participants with plantar fasciitis, would the application of a myofascial release treatment for 15 minutes have equivalent effects to myofascial release applied for 30 minutes, in the pain and stiffness of the gastrocnemius muscle?

ELIGIBILITY:
Inclusion Criteria:

* Study participants must be diagnosed with PF
* Age between 18 to 60 years a clinical diagnosis of unilateral PF according to the clinical practice guidelines of the orthopedic section of the American Physical Therapy Association (APTA).
* Pain intensity > 2 on the numerical pain rating scale (NPRS).
* Pain that is most intense upon awakening and decreases during walking. • Duration of pain greater than 3 months and less than 7 months.
* Both sexes.

Exclusion Criteria:

* Who have received ankle or foot interventions within the previous three months, such as physical therapy (manual therapy, exercise, physical agents), injections, long-term history of steroid use.
* History of surgery on the ankle, foot, or inner leg.
* Other causes of heel pain: arthritic (fibromyalgia, gout, rheumatoid arthritis, seronegative spondyloarthropathies), infectious (diabetic ulcers, osteomyelitis, plantar warts), neurological (lumbar radiculopathy (L4-S2), nerve entrapment (branches of posterior tibial nerve), neuroma, tarsal tunnel syndrome, (posterior tibial nerve), trauma (calcaneal stress fracture), tumor (Ewing's sarcoma, neuroma), vascular and pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Morning pain intensity measured with the Numeric Pain Rating Scale (NPRS) | It will be measured at Baseline, up to 15 min after the first session, at 4 weeks and at 4 weeks after the end of the treatment
  The Numeric Pain Rating Scale (NPRS) measures pain intensity from 0 to 11 points (0, no pain; 10, worst pain imaginable).(18) Numeric pain scales have been shown to be reliable and valid.(25) In addition, the DCMI (minimally clinically important difference) has been reported to be 2 points.(26)

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | It will be measured at Baseline, up to 15 min after the first session, at 4 weeks and at 4 weeks after the end of the treatment
  The pressure pain threshold (PPT), defined as the minimum pressure to induce a change from a pressure sensation to a pain sensation.(27) The score is obtained from the average of 3 repeated measurements, with a 30 second rest between each one, a method that has demonstrated validity and high reliability with ICC=0.91 (95% CI: 0.82, 0.97).(19, 28) The PPT will be evaluated with an Algometer (Wagner Instruments FPX 50). The pressure (force divided by the surface area) will be applied at a speed of approximately 1kg/cm2/s. It will be measured on the most sensitive point of the lower surface of the calcaneus, posterior surface of the calcaneus, soleus muscle and internal and lateral gastrocnemius muscle.(13, 29) To measure each of these points, the subject must be placed face down on the stretcher, with the extremity to be evaluated uncovered.
Calf muscle stiffness (Silfverskiöl test) | It will be measured at Baseline, up to 15 min after the first session, at 4 weeks and at 4 weeks after the end of the treatment
  Gastrocnemius stiffness or tightness will be assessed with the Silfverskiöld test.(20)The measurement explores the degree of passive dorsiflexion of the ankle in the supine position (with a goniometer), in two positions: with the knee extended and flexed (90°), where the hindfoot is in a neutral or varus position. A moderate force load is applied under the forefoot (it is recommended to apply the goniometric measurement with a force between 1.7 and 2kg),(30) the expected difference for the test to be positive is a minimum of 13 degrees of difference.(20) The reliability at the intra-evaluator level with ICC (95% CI) that fluctuates between 0.845 to 0.924.(31) A digital goniometer will be used (brand: baseline evaluation instruments; model: 12-1027; company: enterprises; Country: USA).
Functionality (Foot Function Index (FFI)) | It will be measured at Baseline, up to 15 min after the first session, at 4 weeks and at 4 weeks after the end of the treatment
  Functionality will be assessed through the Foot Function Index (FFI), recommended for subjects who suffer from heel pain,(5) and validated in Spanish.(21) It is a self-administered index consisting of 23 items that measure pain, disability and activity restriction, which has been shown to be reliable, valid and sensitive to foot alterations.(34-36)
Health-related quality of life (SF-12) | It will be measured at Baseline, at 4 weeks and at 4 weeks after the end of the treatment
  Health-related quality of life will be assessed with the SF-12 health questionnaire, which is a shortened version of the SF-36. This scale has 12 items with Likert-style response opinions (3 to 6 points) and a dichotomous scale, it has two summary components, physical (PCS) and mental (MCS), and it summarizes 8 dimensions: physical function, physical role, bodily pain, general health, vitality, social function, emotional role and mental health. The maximum score of the survey indicates good quality of life and is valid in Spanish (correlation with back pain PCS-12 (r= -0.405, P<0.001) and MCS-12 (r=-0.326, P=0.0001)) and reliable (Cronbach's alpha coefficient PCS-12 was 0.77 and MCS-12 was 0.8), in patients with musculoskeletal pain.
Perception of change (Patient Global Impression of Change) | It will be measured at at 4 weeks and at 4 weeks after the end of the treatment
  Satisfaction after the intervention is measured through the perception of change after the intervention, applying the scale "Patient Global Impression of Change" (PGIC). The results will reflect the patient's belief about the effect of the applied treatment. (22) The scale consists of a 7-point verbal scale, with the options "I have improved a lot", "I have improved quite a bit", "I have improved a little", "I am the same", "I have worsened a little", "I have worsened quite a bit" and "I have worsened a lot". (37, 38) A clinically significant improvement is considered to be achieved when the items "I have improved a lot", "I have improved quite a bit" are scored. The test-retest reliability of the global rating of the change scales is excellent (ICC=0.90). (39)
Foot health (Foot Health Status Questionnaire (FHSQ) | It will be measured at Baseline, at 4 weeks and at 4 weeks after the end of the treatment
  Foot health will be measured with the "Foot Health Status Questionnaire (FHSQ)" questionnaire, this scale is validated in Spanish. (24) In addition, it has been shown to have content validity, construct validity, reliability and good responsiveness in patients with plantar fasciitis, who were users of orthopedic physiotherapy.(40)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Laboratory, Department of Physical Therapy, Faculty of Health Sciences, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
The demographic characteristics and the data regarding the main variable and the secondary variables of the participants will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available indefinitely from the moment the results are published.
Access Criteria: Data will be available upon request to the principal investigator or the corresponding author of related publications

REFERENCES:
- [Background] Kinney AR, Eakman AM, Graham JE. Novel Effect Size Interpretation Guidelines and an Evaluation of Statistical Power in Rehabilitation Research. Arch Phys Med Rehabil. 2020 Dec;101(12):2219-2226. doi: 10.1016/j.apmr.2020.02.017. Epub 2020 Apr 6. PMID 32272106
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences: L. Erlbaum Associates; 1988.
- [Background] Flight L, Julious SA. Practical guide to sample size calculations: non-inferiority and equivalence trials. Pharm Stat. 2016 Jan-Feb;15(1):80-9. doi: 10.1002/pst.1716. Epub 2015 Nov 25. PMID 26604186
- [Background] Martin RL, Irrgang JJ. A survey of self-reported outcome instruments for the foot and ankle. J Orthop Sports Phys Ther. 2007 Feb;37(2):72-84. doi: 10.2519/jospt.2007.2403. PMID 17366962
- [Background] Kamper D, Barin K, Parnianpour M, Reger S, Weed H. Preliminary investigation of the lateral postural stability of spinal cord-injured individuals subjected to dynamic perturbations. Spinal Cord. 1999 Jan;37(1):40-6. doi: 10.1038/sj.sc.3100747. PMID 10025694
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Angst F, Aeschlimann A, Stucki G. Smallest detectable and minimal clinically important differences of rehabilitation intervention with their implications for required sample sizes using WOMAC and SF-36 quality of life measurement instruments in patients with osteoarthritis of the lower extremities. Arthritis Rheum. 2001 Aug;45(4):384-91. doi: 10.1002/1529-0131(200108)45:43.0.CO;2-0. PMID 11501727
- [Background] Budiman-Mak E, Conrad KJ, Mazza J, Stuck RM. A review of the foot function index and the foot function index - revised. J Foot Ankle Res. 2013 Feb 1;6(1):5. doi: 10.1186/1757-1146-6-5. PMID 23369667
- [Background] Saag KG, Saltzman CL, Brown CK, Budiman-Mak E. The Foot Function Index for measuring rheumatoid arthritis pain: evaluating side-to-side reliability. Foot Ankle Int. 1996 Aug;17(8):506-10. doi: 10.1177/107110079601700814. PMID 8863033
- [Background] Budiman-Mak E, Conrad KJ, Roach KE. The Foot Function Index: a measure of foot pain and disability. J Clin Epidemiol. 1991;44(6):561-70. doi: 10.1016/0895-4356(91)90220-4. PMID 2037861
- [Background] Luo X, George ML, Kakouras I, Edwards CL, Pietrobon R, Richardson W, Hey L. Reliability, validity, and responsiveness of the short form 12-item survey (SF-12) in patients with back pain. Spine (Phila Pa 1976). 2003 Aug 1;28(15):1739-45. doi: 10.1097/01.BRS.0000083169.58671.96. PMID 12897502
- [Background] Schmidt S, Vilagut G, Garin O, Cunillera O, Tresserras R, Brugulat P, Mompart A, Medina A, Ferrer M, Alonso J. [Reference guidelines for the 12-Item Short-Form Health Survey version 2 based on the Catalan general population]. Med Clin (Barc). 2012 Dec 8;139(14):613-25. doi: 10.1016/j.medcli.2011.10.024. Epub 2012 Jan 11. Spanish. PMID 22244683
- [Background] DiGiovanni CW, Kuo R, Tejwani N, Price R, Hansen ST Jr, Cziernecki J, Sangeorzan BJ. Isolated gastrocnemius tightness. J Bone Joint Surg Am. 2002 Jun;84(6):962-70. doi: 10.2106/00004623-200206000-00010. PMID 12063330
- [Background] AlKhadhrawi N, Alshami A. Effects of myofascial trigger point dry cupping on pain and function in patients with plantar heel pain: A randomized controlled trial. J Bodyw Mov Ther. 2019 Jul;23(3):532-538. doi: 10.1016/j.jbmt.2019.05.016. Epub 2019 May 23. PMID 31563366
- [Background] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Background] Vanderweeen L, Oostendorp RA, Vaes P, Duquet W. Pressure algometry in manual therapy. Man Ther. 1996 Dec;1(5):258-265. doi: 10.1054/math.1996.0276. PMID 11440515
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653
- [Background] Dominguez-Munoz FJ, Garcia-Gordillo MA, Diaz-Torres RA, Hernandez-Mocholi MA, Villafaina S, Collado-Mateo D, Jimenez-Fernandez C, Igual-Fraile D, Perez-Escanilla F, Martin-Gomez G, Adsuar JC, Gusi N. Foot Health Status Questionnaire (FHSQ) in Spanish People with Type 2 Diabetes Mellitus: Preliminary Values Study. Int J Environ Res Public Health. 2020 May 22;17(10):3643. doi: 10.3390/ijerph17103643. PMID 32455874
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Paez-Moguer J, Budiman-Mak E, Cuesta-Vargas AI. Cross-cultural adaptation and validation of the Foot Function Index to Spanish. Foot Ankle Surg. 2014 Mar;20(1):34-9. doi: 10.1016/j.fas.2013.09.005. Epub 2013 Nov 16. PMID 24480497
- [Background] Barouk P, Barouk LS. Clinical diagnosis of gastrocnemius tightness. Foot Ankle Clin. 2014 Dec;19(4):659-67. doi: 10.1016/j.fcl.2014.08.004. Epub 2014 Sep 26. PMID 25456715
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Jensen MP, Turner JA, Romano JM. What is the maximum number of levels needed in pain intensity measurement? Pain. 1994 Sep;58(3):387-392. doi: 10.1016/0304-3959(94)90133-3. PMID 7838588
- [Background] Sheldon A, Karas S. Adverse events associated with manual therapy of peripheral joints: A scoping review. J Bodyw Mov Ther. 2022 Jul;31:159-163. doi: 10.1016/j.jbmt.2022.04.012. Epub 2022 Apr 20. PMID 35710214
- [Background] Tu P. Heel Pain: Diagnosis and Management. Am Fam Physician. 2018 Jan 15;97(2):86-93. PMID 29365222
- [Background] McClinton SM, Cleland JA, Flynn TW. Predictors of response to physical therapy intervention for plantar heel pain. Foot Ankle Int. 2015 Apr;36(4):408-16. doi: 10.1177/1071100714558508. Epub 2014 Nov 3. PMID 25367253
- [Background] Shashua A, Flechter S, Avidan L, Ofir D, Melayev A, Kalichman L. The effect of additional ankle and midfoot mobilizations on plantar fasciitis: a randomized controlled trial. J Orthop Sports Phys Ther. 2015 Apr;45(4):265-72. doi: 10.2519/jospt.2015.5155. Epub 2015 Mar 4. PMID 25739844
- [Background] Jones B, Jarvis P, Lewis JA, Ebbutt AF. Trials to assess equivalence: the importance of rigorous methods. BMJ. 1996 Jul 6;313(7048):36-9. doi: 10.1136/bmj.313.7048.36. PMID 8664772
- [Background] Fuentes C J, Armijo-Olivo S, Magee DJ, Gross DP. A preliminary investigation into the effects of active interferential current therapy and placebo on pressure pain sensitivity: a random crossover placebo controlled study. Physiotherapy. 2011 Dec;97(4):291-301. doi: 10.1016/j.physio.2011.01.001. Epub 2011 Feb 5. PMID 22051585
- [Background] Ajimsha MS, Binsu D, Chithra S. Effectiveness of myofascial release in the management of plantar heel pain: a randomized controlled trial. Foot (Edinb). 2014 Jun;24(2):66-71. doi: 10.1016/j.foot.2014.03.005. Epub 2014 Mar 21. PMID 24703512
- [Background] Saban B, Deutscher D, Ziv T. Deep massage to posterior calf muscles in combination with neural mobilization exercises as a treatment for heel pain: a pilot randomized clinical trial. Man Ther. 2014 Apr;19(2):102-8. doi: 10.1016/j.math.2013.08.001. Epub 2013 Sep 3. PMID 24090993
- [Background] Mischke JJ, Jayaseelan DJ, Sault JD, Emerson Kavchak AJ. The symptomatic and functional effects of manual physical therapy on plantar heel pain: a systematic review. J Man Manip Ther. 2017 Feb;25(1):3-10. doi: 10.1080/10669817.2015.1106818. Epub 2016 Apr 26. PMID 28855787
- [Background] Fraser JJ, Corbett R, Donner C, Hertel J. Does manual therapy improve pain and function in patients with plantar fasciitis? A systematic review. J Man Manip Ther. 2018 May;26(2):55-65. doi: 10.1080/10669817.2017.1322736. Epub 2017 May 3. PMID 29686479
- [Background] McKenney K, Elder AS, Elder C, Hutchins A. Myofascial release as a treatment for orthopaedic conditions: a systematic review. J Athl Train. 2013 Jul-Aug;48(4):522-7. doi: 10.4085/1062-6050-48.3.17. Epub 2013 Apr 3. PMID 23725488
- [Background] Martin RL, Davenport TE, Reischl SF, McPoil TG, Matheson JW, Wukich DK, McDonough CM; American Physical Therapy Association. Heel pain-plantar fasciitis: revision 2014. J Orthop Sports Phys Ther. 2014 Nov;44(11):A1-33. doi: 10.2519/jospt.2014.0303. PMID 25361863
- [Background] Rhim HC, Kwon J, Park J, Borg-Stein J, Tenforde AS. A Systematic Review of Systematic Reviews on the Epidemiology, Evaluation, and Treatment of Plantar Fasciitis. Life (Basel). 2021 Nov 24;11(12):1287. doi: 10.3390/life11121287. PMID 34947818
- [Background] Thomas MJ, Whittle R, Menz HB, Rathod-Mistry T, Marshall M, Roddy E. Plantar heel pain in middle-aged and older adults: population prevalence, associations with health status and lifestyle factors, and frequency of healthcare use. BMC Musculoskelet Disord. 2019 Jul 20;20(1):337. doi: 10.1186/s12891-019-2718-6. PMID 31325954
- [Background] Hill CL, Gill TK, Menz HB, Taylor AW. Prevalence and correlates of foot pain in a population-based study: the North West Adelaide health study. J Foot Ankle Res. 2008 Jul 28;1(1):2. doi: 10.1186/1757-1146-1-2. PMID 18822153